CLINICAL TRIAL: NCT03003221
Title: Improving Dental Care and Oral Health in Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Massachusetts General Hospital (Other); Nationwide Children's Hospital (Other); California State University, Fullerton (Other); Healthy Smiles for Kids of Orange County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-3043
Record Dates: First submitted 2016-12-20; First posted 2016-12-26 (Estimated); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Autism Spectrum Disorder
Keywords: Parent training; Dental care
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- AIR-P Dental Toolkit (Active Comparator): Families will be provided with the Autism Intervention Research Network on Physical Health (AIR-P) Dental Toolkit.
  Interventions: Behavioral: AIR-P Dental Toolkit
- Parent Training (Experimental): Families randomized to the Parent Training condition will be provided with the AIR-P Dental Toolkit and a 10-week behavioral parent-training intervention with additional booster sessions.
  Interventions: Behavioral: AIR-P Dental Toolkit; Behavioral: Parent Training

INTERVENTIONS:
Behavioral: AIR-P Dental Toolkit — The AIR-P Dental Toolkit is designed to provide caregivers with guidance and information related to dental care and support strategies for children with autism spectrum disorder.
Behavioral: Parent Training — The parent-training intervention integrates strategies shown to be efficacious for: 1) improving adherence to dental care, 2) enhancing dental experiences for children with neurotypical development and high levels of dental fear, and 3) evidence-based behavioral techniques established for children with autism spectrum disorder.
  Arms: Parent Training

SUMMARY:
A randomized controlled trial (at sites) comparing the efficacy of the established AIR-P Dental Toolkit (control condition) to a combined regimen involving the Dental Toolkit and parent-mediated behavioral intervention (intervention condition) to improve home dental care, oral health outcomes, and dental office visit experiences.

DETAILED DESCRIPTION:
Participation in routine dental care is a significant challenge for children with autism spectrum disorder (ASD) due to a variety of factors, including considerations related to ASD symptoms and associated anxiety and behavioral difficulties. Lack of routine, effective dental care has contributed to a substantial unmet healthcare need for children with ASD, who are at increased risk for excessive plaque, caries, and oral infections.

The purpose of this study is to test a parent-training intervention designed to improve home dental hygiene, compliance with dental office visits, and oral health outcomes in children with autism spectrum disorder. Families of children with an existing diagnosis of ASD will be recruited for participation. All families will receive the Autism Intervention Research Network on Physical Health (AIR-P) Dental Toolkit, which is designed to provide parents with guidance and information about dental care and support strategies for children with ASD. Some families will also participate in a 10-week behavioral parent-training intervention focused on improving home dental care and dental office visit experiences.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking families of children ages 3 to 13 years and 11 months.
* Current diagnosis of ASD confirmed by baseline assessment.
* Parent-reported difficulty participating in dental care.
* Confirmed absence of dental screenings or exams/visits within the previous 6 months.
* Underserved status as defined by Medicaid eligibility.

Exclusion Criteria:

* Children who present with an acute dental condition requiring emergency treatment.
* Children who are currently taking, or have recently discontinued, medications that affect oral and gingival health.
* Anything that, in the opinion of the Site Principal Investigator, would place the subject at unwarranted risk or materially reduce their contribution to the trial's aims due to inability or refusal to adhere to trial procedures and follow-up.

Families will be asked to refrain from participating in any non-study adaptive behavior interventions or therapies focused on dental hygiene. Families will also be asked not to participate in any non-study dental screenings or exams for the duration of the investigation.

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 119 (Actual)
Dates: Start 2016-12; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Frequency of tooth brushing at home | Change from Baseline frequency of tooth brushing at 6 months
  Parent-reported frequency of successful (twice-daily) child tooth brushing completed at home during the past week.
Child oral health according to standardized measures from visual exam | Change from Baseline child oral health at 6 months
  Dentist ratings of child oral health according to standardized measures from visual exam.

SECONDARY OUTCOMES:
Child behavior during tooth brushing at home according to questionnaire | Change from Baseline child behavior at 6 months
  Parent-reported child behavioral compliance with home dental hygiene during past week according to questionnaire.
Observed child anxiety and behavior at the dental office visit as indexed by observer ratings on the Venham Anxiety and Behavior Scales (aggregate composite) | Change from Baseline anxiety and behavior at 6 months
  Child compliance with dental visit as indexed by observer ratings on the Venham Anxiety and Behavior Scales (aggregate composite).
Dentist-reported child behavioral compliance during dental office visit as indexed by questionnaire | Change from Baseline behavioral compliance at 6 months
  Dentist-reported child behavioral compliance with dental visit as indexed by questionnaire.
Completion of dental visit procedures according to questionnaire | Change from Baseline completion of dental visit procedures at 6 months
  Dentist-reported completion of visit procedures according to questionnaire.

OTHER OUTCOMES:
Parenting Stress according to questionnaire | Change from Baseline parent-reported parenting stress at 6 months
  Parent-reported parenting stress according to questionnaire.
Perceived Parenting Competence according to questionnaire | Change from Baseline parent-reported perceived parenting competence at 6 months
  Parent-reported perceived parenting competence according to questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Steinberg-Epstein, MD, Study Chair — University of California, Irvine; Rachel M Fenning, PhD, Principal Investigator — University of California-Irvine; California State University-Fullerton; Eric Butter, PhD, Principal Investigator — Nationwide Children's Hospital
Locations (2):
- United States (2):
  - University of California Irvine, Irvine, California
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD data beyond collaborating sites (MGH and NCH).

REFERENCES:
- [Derived] Fenning RM, Butter EM, Macklin EA, Norris M, Hammersmith KJ, McKinnon-Bermingham K, Chan J, Stephenson KG, Albright C, Scherr J, Moffitt JM, Lu F, Spaulding R, Guijon J, Hess A, Coury DL, Kuhlthau KA, Steinberg-Epstein R. Parent Training for Dental Care in Underserved Children With Autism: A Randomized Controlled Trial. Pediatrics. 2022 May 1;149(5):e2021050691. doi: 10.1542/peds.2021-050691. PMID 35211746